CLINICAL TRIAL: NCT04185246
Title: A Multicenter, Open-Label, Dose Ascending Study to Evaluate the Safety of NH002 as a Contrast Agent in Cardiac Echocardiography
Brief Title: A Dose Ascending Study to Evaluate the Safety of NH002 as a Contrast Agent in Cardiac Echocardiography
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Trust Bio-sonics, Inc. (Industry)
Collaborators: StatPlus,Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NH002-LV
Record Dates: First submitted 2019-11-06; First posted 2019-12-04 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Disease
Keywords: Echo; Echocardiogram; Cardiac ultrasound; suboptimal; contrast agent; enhancing agent; LVO; LVEBD
MeSH Terms: conditions — Heart Diseases | interventions — Echocardiography

STUDY DESIGN:
Masking Description: The reviewer of echocardiograms in this trial is blinded to the treatment assignments and subject identifiers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Subjects will be enrolled with sequential allocation to 1 of 3 cohorts with the following intravenous (IV) doses of NH002: 2.5 µl/kg, 5.0 µl/kg, or 10.0 µl/kg.
  Each patient will undergo an unenhanced ultrasound examination and a NH002 contrast-enhanced examination on the same day
  Interventions: Drug: NH002 (Perflutren Lipid Microspheres) Injectable Suspension; Diagnostic Test: Echocardiogram

INTERVENTIONS:
Drug: NH002 (Perflutren Lipid Microspheres) Injectable Suspension — NH002 is formulated as a microbubble injectable suspension for intravenous administration. NH002 requires an activation process prior to use.
Diagnostic Test: Echocardiogram — Each patient will undergo an unenhanced ultrasound examination and a NH002 contrast-enhanced examination on the same day.

SUMMARY:
NH002 (Perflutren Lipid Microspheres) Injectable Suspension is an ultrasound contrast agent for use in patients with suboptimal echocardiograms to opacify the left ventricular (LV) chamber and to improve the delineation of the LV endocardial border. The primary objective of this study is to evaluate the safety and tolerability of 3 ascending doses of NH002.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 20 years of age or older
2. Ability to understand and the willingness to provide written informed consent
3. Suspected of having cardiac disease or undergoing evaluation of cardiac anatomy for congenital heart disease
4. Negative pregnancy test within 24 hours of the procedure if subject is a woman of childbearing potential

Exclusion Criteria:

1. Known right-to-left, bidirectional, or transient right-to-left cardiac shunt(s)
2. Chronic obstructive pulmonary disease
3. Ejection fraction at screening or baseline <40%
4. Uncontrolled serious ventricular arrhythmias or at high risk for arrhythmias due to prolongation of the QT interval (QT corrected by Fridericia's formula >450 msec in males and >470 msec in females)
5. Clinically significant abnormality in renal and liver function tests (alanine aminotransferase/aspartate aminotransferase >2 × upper limit of normal [ULN]; serum creatinine > 1.5 × ULN)
6. Known or suspected hypersensitivity to one or more of the ingredients of NH002, perflutren, or other echocardiographic contrast agent
7. Received an investigational compound within 30 days before enrolling in the study
8. Received any contrast agent either intravascularly or orally within 48 hours before NH002 administration
9. Pregnant or lactating female (conception during the study should be avoided)
10. Serious medical or psychiatric illness/condition likely, in the judgment of the investigator, to interfere with compliance to protocol treatment/research
11. Clinically unstable cardiopulmonary conditions considered not suitable for participation in the trial, in the judgment of the investigator
12. Uncontrolled arterial hypertension (defined as systolic blood pressure ≥ 200 mmHg or diastolic blood pressure ≥ 110 mmHg) or arterial hypotension (defined as systolic blood pressure ≤ 90 mmHg)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chung Yu, Principal Investigator — Taipei Veterans General Hospital, Taiwan; Chung-Lieh Hung, Principal Investigator — Taipei Mackay Memorial Hospital
Locations (2):
- Taiwan (2):
  - Taipei Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Subjects will be enrolled with the following intravenous (IV) doses of NH002: 2.5 µl/kg.
  Each patient will undergo an unenhanced ultrasound examination and a NH002 contrast-enhanced examination on the same day
- Cohort 2: Subjects will be enrolled with the following intravenous (IV) doses of NH002: 5.0 µl/kg.
  Each patient will undergo an unenhanced ultrasound examination and a NH002 contrast-enhanced examination on the same day
- Cohort 3: Subjects will be enrolled with the following intravenous (IV) doses of NH002: 10.0 µl/kg.
  Each patient will undergo an unenhanced ultrasound examination and a NH002 contrast-enhanced examination on the same day
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Participants received single intravenous bolus injection dose of NH002 2.5 µl/kg.
- Cohort 2: Participants received single intravenous bolus injection dose of NH002 5.0 µl/kg.
- Cohort 3: Participants received single intravenous bolus injection dose of NH002 10.0 µl/kg.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (14.77) | 38.8 (10.29) | 36.8 (11.42) | 39.7 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 6 | 17
  Male | 8 | 5 | 6 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 12 | 12 | 12 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeter] | 168.4 (11.396) | 163.7 (10.93) | 166.74 (11.991) | 166.28 (11.29)
Weight [Mean (Standard Deviation); unit: kilogram] | 76.88 (21.992) | 63.17 (13.131) | 73.59 (22.279) | 71.21 (19.933)

OUTCOME MEASURES:

1. Primary Outcome: 12-lead ECGs
Description: Standard 12-lead ECGs will be assessed from pre-injection to 60 minutes post-injection for changes in QT/ corrected QT(QTc) interval (in ms) and ECG morphology; each standard 12-lead ECG assessment will be scored as either normal or abnormal
Time Frame: From pre-injection to 60 minutes post injection
Population: All abnormal findings of 12-lead ECG interpretations after dosing were assessed as non-clinically significant and not related to NH002.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 12 | 12
millisecond
  Baseline (QT) | 393.9 (19.37) | 392.0 (24.07) | 386.3 (25.99)
  Change of Baseline (QT) at 10 minutes post-dose | 2.8 (13.65) | -6.0 (13.16) | 6.8 (17.65)
  Change of Baseline (QT) at 30 minutes post-dose | 10.8 (13.28) | 6.0 (12.59) | 16.0 (13.4)
  Change of Baseline (QT) at 60 minutes post-dose | 7.1 (17.17) | 3.4 (17.17) | 10.6 (9.59)
  Baseline (QTc) | 415.1 (21.71) | 415.9 (20.38) | 404.6 (15.32)
  Change of baseline (QTc) at 10 minutes post-dose | 1.3 (13.92) | -6.4 (10.95) | 7.8 (7.7)
  Change of baseline (QTc) at 30 minutes post-dose | 0.4 (14.25) | -1.3 (12.14) | 8.8 (9.17)
  Change of baseline (QTc) at 60 minutes post-dose | -0.1 (13.03) | -3.0 (11.96) | 6.9 (5.88)

2. Primary Outcome: Body Temperature
Description: Monitor for any changes in body temperature (in Celsius degree)
Time Frame: From pre-injection to 120 minutes post injection
Measure: Mean (Standard Deviation); unit: Celsius degree
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 12 | 12
Celsius degree
  Baseline | 36.76 (0.294) | 36.73 (0.306) | 36.76 (0.385)
  Change from baseline at 5 minutes post-dose | -0.01 (0.215) | -0.02 (0.195) | -0.01 (0.268)
  Change from baseline at 10 minutes post-dose | -0.01 (0.312) | 0.07 (0.235) | -0.06 (0.207)
  Change from baseline at 30 minutes post-dose | -0.07 (0.328) | 0.11 (0.215) | 0 (0.2)
  Change from baseline at 60 minutes post-dose | -0.08 (0.457) | 0.05 (0.271) | -0.18 (0.313)
  Change from baseline at 120 minutes post-dose | -0.07 (0.442) | 0.1 (0.283) | -0.02 (0.518)

3. Primary Outcome: Heart Rate
Description: Monitor for any changes in heart rate (in beats/min)
Time Frame: From pre-injection to 120 minutes post injection
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 12 | 12
beats/minute
  Baseline | 70.1 (9.93) | 71.3 (7.73) | 69.0 (8.06)
  Change from baseline at 10 minutes post-dose | -0.7 (2.71) | -0.1 (5.87) | -0.1 (3.73)
  Change from baseline at 30 minutes post-dose | -3.0 (5.34) | -1.3 (5.99) | -0.3 (6.85)
  Change from baseline at 60 minutes post-dose | -0.9 (5.96) | -1.2 (4.37) | 0.7 (4.56)
  Change from baseline at 120 minutes post-dose | 4.9 (10.29) | 6.8 (12.4) | 8.3 (9.9)

4. Primary Outcome: Respiratory Rate
Description: Monitor for any changes in respiratory rate (in breaths/min)
Time Frame: From pre-injection to 120 minutes post injection
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 12 | 12
breaths/minute
  Baseline | 15.6 (3.55) | 15.1 (2.07) | 16.9 (4.44)
  Change from baseline at 10 minutes post-dose | 0.6 (3.8) | -0.6 (3.29) | -1.4 (3.12)
  Change from baseline at 30 minutes post-dose | 0.9 (3.09) | -0.8 (3.28) | -1.3 (4.71)
  Change from baseline at 60 minutes post-dose | 0.5 (3.85) | -0.9 (2.75) | -2.3 (4.09)
  Change from baseline at 120 minutes post-dose | 0.8 (3.43) | -0.5 (3.61) | -1.3 (4.48)

5. Primary Outcome: Blood Pressure
Description: Monitor for any changes in blood pressure (in mmHg)
Time Frame: From pre-injection to 120 minutes post injection
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 12 | 12
mmHg
  Baseline (SBP) | 132.8 (14.93) | 106.8 (15.6) | 112.7 (16.33)
  Change from baseline (SBP) at 10 minutes post-dose | -2.5 (9.48) | 0.5 (6.45) | -0.3 (7.76)
  Change from baseline (SBP) at 30 minutes post-dose | -5.2 (11.54) | 4.8 (13.33) | 4.1 (9.46)
  Change from baseline (SBP) at 60 minutes post-dose | -4.8 (15.03) | 1.5 (12.59) | 6.0 (10.44)
  Change from baseline (SBP) at 120 minutes post-dose | -4.0 (13.1) | 7.6 (15.47) | 13.8 (19.6)
  Baseline (DBP) | 85.2 (11.61) | 68.5 (13.3) | 71.5 (11.76)
  Change from baseline (DBP) at 10 minutes post-dose | -2.6 (6.56) | 0 (4.92) | 2.6 (5.96)
  Change from baseline (DBP) at 30 minutes post-dose | -3.9 (8.12) | 4.1 (10.66) | 3.1 (9.6)
  Change from baseline (DBP) at 60 minutes post-dose | -3.0 (10.4) | 3.6 (11.52) | 7.8 (11.58)
  Change from baseline (DBP) at 120 minutes post-dose | -2.3 (7.94) | 6.8 (14.16) | 8.7 (14.5)

6. Primary Outcome: Thrombin Time (TT) and Activated Partial Thromboplastin Time (aPTT)
Description: Monitor for any changes in TT and aPTT
Time Frame: From pre-injection to 240 minutes post-injection
Population: The total number of subjects in cohort 2 who underwent TT testing was 11.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 12 | 12
seconds
  Baseline (TT) | 18.6 (3.145) | 17.81 (0.667) | 16.7 (1.836)
  Change from baseline (TT) at 60 minutes post-dose | 0.22 (0.395) | -0.12 (0.387) | -0.24 (0.724)
  Change from baseline (TT) at 120 minutes post-dose | 0.06 (0.528) | 0.05 (0.95) | -0.3 (0.662)
  Change from baseline (TT) at 240 minutes post-dose | 0.11 (0.497) | -0.05 (0.62) | 0.31 (1.274)
  Baseline (APTT) | 31.54 (3.888) | 28.76 (27.81) | 28.87 (2.796)
  Change from baseline (APTT) at 60 minutes post-dose | -0.3 (2.625) | -1.05 (2.184) | -0.8 (2.921)
  Change from baseline (APTT) at 120 minutes post-dose | -0.49 (3.11) | -0.48 (1.788) | -0.61 (2.586)
  Change from baseline (APTT) at 240 minutes post-dose | -0.55 (3.191) | -0.68 (1.516) | -1.5 (2.375)

7. Primary Outcome: Cardiac Troponin I
Description: Monitor for any changes in Cardiac troponin I
Time Frame: pre-injection and 240 minutes post-injection
Population: Troponin I was utilized at site 102. The sample sizes were 5, 7, and 7 for cohorts 1, 2, and 3, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 7 | 7
ng/mL
  Baseline (troponin I) | 0.005 (0.000) | 0.005 (0.000) | 0.005 (0.000)
  240 minutes after dosing (troponin I) | 0.005 (0.000) | 0.005 (0.000) | 0.005 (0.000)
  Change from baseline (troponin I) at 240 minutes post-dose | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)

8. Primary Outcome: Oxygen Saturation by Pulse Oximetry (SpO2)
Description: Monitor for any changes in SpO2
Time Frame: From pre-injection to 120 minutes post-injection
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 12 | 12
percentage
  Baseline | 98.8 (1.06) | 98.9 (1.51) | 98.3 (1.14)
  Change from baseline at 10 minutes post-dose | 0.4 (1.31) | 0.3 (0.62) | -0.4 (1.38)
  Change from baseline at 30 minutes post-dose | 0.2 (1.27) | 0.3 (1.29) | -0.3 (0.87)
  Change from baseline at 60 minutes post-dose | 0.5 (1.88) | 0.4 (1.38) | 0.8 (1.22)
  Change from baseline at 120 minutes post-dose | 0 (1.13) | -0.2 (1.64) | 0.2 (0.94)

9. Primary Outcome: Rate of Any Potential Adverse Allergic Reaction
Description: Monitor for any potential adverse allergic reaction
Time Frame: From pre-injection to 240 minutes post-injection
Population: One subject allergic to the tap (not injection site) at 120 minutes after dosing. It was determined that there was no relationship between the data and the IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

10. Secondary Outcome: Left Ventricular Opacification (LVO)
Description: The percentage of subjects with moderate or complete left ventricular opacification (LVO), defined by an LVO grade of 2 (moderate) or 3 (complete), as assessed by the blinded central reader(s).
  The percentage of subjects with complete LVO, defined by an LVO grade of 3 (complete), as assessed by the blinded central reader(s)
Time Frame: Image data obtained pre-injection and within 10 minutes post-injection
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 12 | 12
Participants
  LVO grade of 2 (moderate) or 3 (complete) | 12 | 12 | 12
  LVO grade of 3 (complete) | 11 | 12 | 12

11. Secondary Outcome: Left Ventricular Endocardial Border Delineation (LVEBD)
Description: The change from baseline on the left ventricular endocardial border delineation (LVEBD) score, defined using a standard 12-segment model, as assessed by the blinded central reader(s). The left ventricular (LV) endocardium of the 4- or 2- chamber apical views are divided into 6 segments, with 2 basal, mid- and apical segments in each view. For each segment, LVEBD is graded as follows: 0= inadequate border (border not visible); 1= sufficient (border barely visible); 2= good (border clearly visible). A total delineation score (0-24) is obtained by adding the scores from the 6 individual segments in each of the 2 views.
  The changes from baseline on LVEBD score of subjects with suboptimal LVEBD at baseline, as defined by 2 or more contiguous segments of 6 segments that cannot be visualized reliably in either the apical 4 and/or the 2-chamber view, as assessed by the blinded central reader(s)
Time Frame: Image data obtained pre-injection and within 10 minutes post-injection
Population: There were 9, 10, and 9 subjects with suboptimal baseline values in cohorts 1, 2, and 3, respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 12 | 12
score on a scale
  LVEBD scores_Baseline (all subjects) | 11.5 (6.75) | 8.9 (4.89) | 9.7 (6.68)
  LVEBD scores_Post-dose (all subjects) | 23.0 (3.46) | 23.8 (0.62) | 23.9 (0.29)
  Change from baseline (all subjects) | 11.5 (7.22) | 14.8 (4.71) | 14.3 (6.59)
  LVEBD scores_Baseline (subjects with suboptimal LVEBD at baseline): number analyzed (Participants) | 9 | 10 | 9
  LVEBD scores_Baseline (subjects with suboptimal LVEBD at baseline) | 8.6 (4.48) | 7.4 (3.72) | 7.8 (6.65)
  LVEBD scores_Post-dose (subjects with suboptimal LVEBD at baseline): number analyzed (Participants) | 9 | 10 | 9
  LVEBD scores_Post-dose (subjects with suboptimal LVEBD at baseline) | 22.7 (4.0) | 23.7 (0.67) | 23.9 (0.33)
  Change from baseline (subjects with suboptimal LVEBD at baseline): number analyzed (Participants) | 9 | 10 | 9
  Change from baseline (subjects with suboptimal LVEBD at baseline) | 14.1 (6.11) | 16.3 (3.56) | 16.1 (6.57)

12. Secondary Outcome: Duration of Clinically Useful Contrast
Description: A duration of clinically useful contrast calculated by measuring the time between the disappearance of shadowing effect (useful effect starts) and the time when moderate or full LV enhancement and contrast enhancement are no longer adequate (useful effect ends), as assessed by the blinded central reader(s)
Time Frame: Image data obtained pre-injection and within 10 minutes post-injection
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 12 | 12
minutes | 7.2 (2.458) | 7.67 (1.684) | 3.59 (1.854)

13. Primary Outcome: Cardiac Troponin T
Description: Monitor for any changes in Cardiac troponin T
Time Frame: pre-injection and 240 minutes post-injection
Population: Troponin T was utilized at site 101. The sample sizes were 7, 5, and 5 for cohorts 1, 2, and 3, respectively.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 7 | 5 | 5
ng/L
  Baseline (troponin T) | 4.07 (2.53) | 1.5 (0.0) | 4.38 (1.824)
  240 minutes after dosing (troponin T) | 5.21 (1.368) | 2.3 (1.105) | 5.72 (4.387)
  Change from baseline (troponin T) at 240 minutes post-dose | 1.14 (1.878) | 0.8 (1.105) | 1.34 (3.833)

ADVERSE EVENTS:
Time Frame: Each subject had to be carefully monitored for the development of any AEs throughout the study from the signing of the informed consent form to 7 days after receipt of the dose of study agent.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 2/12 | 7/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=12) | Cohort 2 (N=12) | Cohort 3 (N=12)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT04185246/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT04185246/SAP_001.pdf